CLINICAL TRIAL: NCT04467892
Title: Comparative Study Between the Uses of High Dose Corticosteroid Therapy for Short Duration Versus Low Dose Corticosteroid for Long Duration in Severe Lung Contusion With ARDS
Brief Title: Low Versus High Corticosteroid Use in Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU-11-20
Record Dates: First submitted 2020-06-06; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Methylprednisolone; methyl prednisolonate; Ventilators, Mechanical

STUDY DESIGN:
Intervention Model Description: Patients who had severe chest trauma with massive lung contusion and admitted to King Abdelaziz specialist hospital between January 2018 and February 2020 in the intensive care unit those who showed the following inclusion criteria of ARDS, respiratory failure due to severe lung contusion complicated by VAP enrolled in our study
Masking Description: patients with COPD respiratory failure, patients with congestive heart failure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): . Group A 120 patients, received high dose (30 mg/kg) methylprednisolone slowly intravenous in 250 ml normal saline every 8 hours for only 4 days
  Interventions: Drug: methylprednisolone; Device: ventilators
- Group B (Active Comparator): group B 120 patients, included received 1 mg/kg/day methylprednisolone divided to three doses given every 8 hours for two weeks.
  Interventions: Drug: Methyl Prednisolonate; Device: ventilators

INTERVENTIONS:
Drug: methylprednisolone — received high dose (30 mg/kg) methylprednisolone slowly intravenous in 250 ml normal saline every 8 hours for only 4 days
  Arms: Group A
Drug: Methyl Prednisolonate — received 1 mg/kg/day methylprednisolone divided to three doses given every 8 hours for two weeks.
  Arms: Group B
Device: ventilators — all patients in both groups will be ventilated with CMV for 2 weeks

SUMMARY:
patients who had >3 on Murray score and >6 on CPIS allocated randomly in two groups 120 patients in each. Group A received 30 mg/kg methyl-prednisolone slowly intravenous in 250 mL normal saline every 8 hours for only 48 hours while group B received 1 mg/kg/day methyl-prednisolone divided to three doses given every 8 hours for two weeks. Duration of the study last 16 days, Morbidity considered if no improvement in any or all clinical parameters of both Murray and CPIS scores and failure of weaning of patients from the ventilator at the studied period.

DETAILED DESCRIPTION:
Adult patients aged >18<65 years, hypercapnia with PH <7.25, hypoxic index less than 200 (PaO2/FIO2), bilateral parenchymatous lung infiltration in the chest Xray. All selected patients received conventional ventilation with protective lung strategy for 3 days with Controlled mechanical ventilation mode (CMV), fraction inspired oxygen (FIO2) of 100%, Positive end expiratory pressure (PEEP) adjusted to achieve target arterial oxygen saturation (SPO2) of >90%. Sedation and pain control done by both midazolam and fentanyl infusion to achieve Richmond Agitation- Sedation Scale (RASS) -2. Protective lung strategy applied and include, head elevation more than 45-degree, daily assessment for both analgesic and sedative dose, early naso-gastric feeding to prevent bacterial translocation and flooding of the blood with gram negative septicemia, usage of the minimal PEEP to maintain SPO2 >90%. Qualitative sputum culture was taken after 3 days from ventilation. After 3 days from the conventional ventilation only 240 patients enrolled in our study. Those who had a Murray score (for diagnosis of ARDS) of >3 and CPIS (clinical pulmonary infection score) (for diagnosis of VAP) > 6. All patients were randomly allocated in 2 groups 120 patients in each. All patients received intravenous antibiotics meropenem 1 gm slowly intravenous every 8 hours for the first 8 days then antibiotics was given according to sputum culture and antibiotics sensitivity. Group A received high dose (30 mg/kg) methylprednisolone slowly intravenous in 250 ml normal saline every 8 hours for only 4 days while group B included received 1 mg/kg/day methylprednisolone divided to three doses given every 8 hours for two weeks. This study conducted for 16 days.

VAP diagnosed in our study by CPIS 6 or more while severity of lung contusion assessed by Murray score 3 or more

ELIGIBILITY:
Inclusion Criteria:

* ventilator associated pneumonia patients

Exclusion Criteria:

* post cardiac arrest

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Number of patients weaned from the ventilators | 2 weeks
  followed by arterial oxygen saturation
Number of patients discharge from ICU | 2 weeks
  number of patients weaned and ready to be discharged from ICU

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
medical doctors and intensivist